CLINICAL TRIAL: NCT03492528
Title: Cardiovascular Outcome of Cancer Patients: The "GMEDICO Cohort"
Acronym: GMEDICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-50; 2017-A03362-51 (Other: N°IDRCB)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Prognosis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiovascular patients treated for a cancer (Experimental)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — blood samples

SUMMARY:
The Mediterranean Group of Cardio-Oncology (GMEDICO) brings together French cardiologists and oncologists who have developed a protocol for the monitoring and cardio-oncological management of patients treated for cancer.

This unique organization makes it possible to envisage the creation of a large cohort from which the incidence and predictive factors of cardiovascular toxicity can be determined.

Primary objective: to determine the cardiovascular prognosis of patients treated for cancer and followed up in cardio-oncology.

Secondary objectives

* To determine the clinical, biological and imaging factors associated with cardiovascular events under cancer treatment, in order to define a risk score including clinical, biological (biomarker) and imaging data.
* To create a biological source for testing other biomarkers and conducting genome-wide association studies and genetic factors associated with cardiovascular events under cancer treatment.

DETAILED DESCRIPTION:
Each patient will be monitored for 5 years. Cardio-oncological follow-up and management within these centers will follow a common protocol established and validated in March 2016 on the basis of international recommendations and summaries of the characteristics produced for each drug. Additional blood samples will be taken for the biobanking. Depending on the case, a small skin biopsy will be carried out to analyze the cardiovascular response of in vitro immunotherapy using a reprogramming model of fibroblasts in hiPSC hiPSC (human induced Pluripotent Stem cells)-cardiomyocytes.

ELIGIBILITY:
Inclusion Criteria:

* All adults referred for specialist cardio-oncology consultations before the initiation of a cancer treatment according to pre-established indications will be eligible.

Exclusion Criteria:

* Failure to provide information that makes it impossible to complete a consultation form or refuse to sign the consent.
* Minor or major patient under guardianship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Dosage of cardiac biomarkers | 5 YEARS
  dosage of troponine

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assiatnce Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Dolladille C, Ederhy S, Allouche S, Dupas Q, Gervais R, Madelaine J, Sassier M, Plane AF, Comoz F, Cohen AA, Thuny FR, Cautela J, Alexandre J. Late cardiac adverse events in patients with cancer treated with immune checkpoint inhibitors. J Immunother Cancer. 2020 Jan;8(1):e000261. doi: 10.1136/jitc-2019-000261. PMID 31988143